CLINICAL TRIAL: NCT03928652
Title: Prospective Study for Prognostic And Predictive Biomarkers of Colorectal Cancer
Brief Title: Prognostic Biomarker for CRC
Acronym: PROMOTE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: Lan2019/4/24
Record Dates: First submitted 2019-04-24; First posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and tumor tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this clinical research project is to explore potential biomarkers and validate the predictive and prognostic value of molecular signature in colorectal cancer.

DETAILED DESCRIPTION:
This is a prospective observational study. Tumor tissue specimens and surgical specimens are obtained from the Sixth Affiliated Hospital, Sun Yat-sen University. The samples are analyzed for biomarkers. The biomarkers are correlated with clinical outcomes (failure-free survival, overall survival, tumor response to treatment (e.g. tumor regression grade for rectal cancer), distant metastasis, recurrence and death).

The aim of the analysis is to explore potential biomarkers and validate the predictive and prognostic value of molecular signature in . This will lead to the definition of risk groups and stratification of patients and will help to precision medicine of colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Colon or rectal cancer diagnosed by endoscopic biopsy histopathology;
2. Complete sample information, including sample number, gender, age and clinical molecular diagnostic information, etc.;
3. Sufficient surgical tissue samples are available for testing;
4. untreated colon or rectal cancer patients;
5. Patient able to understand and sign written informed consent
6. No evidence of distant metastasis (M0)

Exclusion Criteria:

1. Previously treated CRC, including cytotoxic drug therapy, targeted drug therapy, etc.;
2. Other malignant tumors;
3. Pregnant women;
4. Hereditary colorectal cancer linked to familial colonic polyposis or Lynch syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly histologically confirmed colorectal cancer and no evidence of distant metastasis
Sampling Method: Probability Sample
Enrollment: 1050 (Estimated)
Dates: Start 2019-04-24 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Failure-free Survival | 3 years
Tumor regression grade | 1 year
  For rectal cancer patients who receive neoadjuvant treatment

SECONDARY OUTCOMES:
Overall survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital, Sun Yet-sen University, Guangzhou, China